CLINICAL TRIAL: NCT00503360
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Masked, 4-Arm Parallel Group Study to Assess the Tolerability, Safety and Efficacy of Two Doses of SAD448 in Subjects With Ocular Hypertension
Brief Title: Tolerability, Safety and Efficacy of SAD448 in Subjects With Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSAD448B2101
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Ocular Hypertension
Keywords: Ocular Hypertension; SAD448
MeSH Terms: conditions — Ocular Hypertension

INTERVENTIONS:
Drug: SAD448

SUMMARY:
This study will evaluate the tolerability and safety of SAD448 and explore the compound's effect on intraocular pressure in subjects with ocular hypertension.

ELIGIBILITY:
Key inclusion criteria:

* Males and females, 18 - 65 years of age, with ocular hypertension
* Females must be post-menopausal or surgically sterile

Key exclusion criteria:

* Diagnosis of glaucoma in either eye
* A history of or current eye conditions or medical problems that would prohibit the use of an investigational drug

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Rates of adverse events and serious adverse events, as well as changes in ophthalmic evaluations, laboratory values, ECGs and vital signs from baseline up to 24 hours post-dosing.

SECONDARY OUTCOMES:
Change in ocular hypertension from baseline up to 24 hours post-dosing. Systemic exposure to SAD448 following the administration of two doses.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative site, Sydney, Australia, Sydney, Australia